CLINICAL TRIAL: NCT04905823
Title: Effect of SARSCoV2 Vaccination in Type 1 Diabetes (CoVaxT1D)
Brief Title: Effect of SARSCoV2 (COVID-19) Vaccination in Type 1 Diabetes (CoVaxT1D)
Acronym: CoVaxT1D
Status: Completed | Type: Observational
Sponsor: Paolo Fiorina, MD (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Sponsor-Investigator, Paolo Fiorina, MD, Professor of Endocrinology, Chief of Endocrinology Division, University of Milan
Organization: University of Milan (Other)
Other Study IDs: CoVaxT1D
Record Dates: First submitted 2021-05-24; First posted 2021-05-28 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 1 diabetes patients: Patients with type 1 diabetes
  Interventions: Diagnostic Test: blood test
- Non-diabetic subjects: Subjects in whom diabetes has not been diagnosed
  Interventions: Diagnostic Test: blood test
- Type 2 diabetes patients: Patients with type 2 diabetes
  Interventions: Diagnostic Test: blood test

INTERVENTIONS:
Diagnostic Test: blood test — assessment of humoral, immune cell response and glycemia

SUMMARY:
Given the high risk of severe SARS-CoV-2 infection, patients with T1D and T2D should represent a priority group to receive the SARS-CoV-2 vaccine. There are currently no studies on diabetic population response to mRNA COVID-19 vaccines. Therefore, in this observational cohort study, investigators will retrospectively analyze the safety and immunogenicity of the mRNA vaccines in eliciting both the humoral and cellular immune response in a subset of patients with T1D who already underwent blood sampling for measuring humoral response against SARSCoV2 for healthcare purposes and based on the clinical practice guidelines. Results will be compared with those obtained in non-diabetic individuals or in patients with non-autoimmune diabetes (T2D).

DETAILED DESCRIPTION:
Since the beginning of the COVID-19 pandemic in March 2020, more than 160 million people have suffered from severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, and more than 3 million deaths occurred. Currently, two vaccines using messenger RNA (mRNA) technology and lipid nanoparticle (LNP) delivery systems have been approved for emergency use by the Food and Drug Administration (FDA) and the European Medicines Agency (EMA): mRNA-1273, Moderna, and BNT162b2, Pfizer. In phase-3 clinical trials, two injections of these vaccines, spaced 21 and 28 days apart, showed efficacy higher than 90% in preventing symptomatic infections. The reported humoral immunity response with the mRNA vaccines was similar to that elicited by convalescent serum obtained from patients who recovered from Covid-19 infection. However, the T-cell mediated reaction to these vaccines remains to be fully elucidated. Diabetic patients are at higher risk of developing severe SARS-CoV-2 infection. In a large observational cohort study, the overall risks of fatal or critical care unit-treated COVID-19 were significantly elevated for patients with diabetes compared with the general population. While patients with Type 2 diabetes (T2D) are usually older and with a higher comorbidity index, the altered immune functions seem to play a major role in patients with Type 1 Diabetes (T1D). Altough an impaired immune response to vaccination was hypothesized in diabetic patients, no evidence has been provided. Given the high risk of severe SARS-CoV-2 infection, patients with T1D and T2D should represent a priority group to receive the COVID-19 vaccine. There are currently no studies on diabetic population response to mRNA COVID-19 vaccines. Therefore, in this observational cohort study, investigators will retrospectively analyze the safety and immunogenicity of the mRNA vaccines in eliciting both the humoral and cellular immune response in a subset of patients with T1D, T2D and in non-diabetic individuals who already underwent blood sampling for measuring humoral response against SARSCoV2 for healthcare purposes and based on the clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria for patients with type 1 diabetes:

* age >16
* History of type 1 diabetes
* previous blood test in search for SARSCoV2 antibodies
* willingness to provide informed consent

Exclusion Criteria for patients with type 1 diabetes:

* age <16 years
* Systemic infections
* Diabetic ketoacidosis in the past 6 weeks
* COVID-19 diagnosis in the previous 6 months

Inclusion Criteria for non-diabetic subjects:

* age >16
* No previous history of diabetes
* previous blood test in search for SARSCoV2 antibodies
* willingness to provide informed consent

Exclusion Criteria for non-diabetic subjects:

* age <16 years
* Systemic infections
* COVID-19 diagnosis in the previous 6 months

Inclusion Criteria for patients with type 2 diabetes:

* age >16
* History of type 2 diabetes but no evidence of autoantibodies
* previous blood test in search for SARSCoV2 antibodies
* willingness to provide informed consent

Exclusion Criteria for patients with type 2 diabetes:

* age <16 years
* Systemic infections
* COVID-19 diagnosis in the previous 6 months

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with T1D, non-diabetic subjects and diabetic patients without T1D (T2D) who underwent blood sampling for testing levels of autoantibodies against SARSCoV2 after SARSCoV2 vaccination will be consecutively included in this retrospective study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | change from baseline number at 2 months
  number of adverse events after SARSCov2 vaccination

SECONDARY OUTCOMES:
Humoral response | change from baseline levels at 2 months
  Levels of antibodies detected against SARSCoV2
Immune cell response | change from baseline levels at 2 months
  T cell response quantification
Values of continuous glucose monitoring | change from baseline values at 2 months
  analysis of glycemic profile measured with continuous glucose monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- ASST FBF-Sacco P.O. Sacco, Milan, MI, Italy

REFERENCES:
- [Derived] D'Addio F, Sabiu G, Usuelli V, Assi E, Abdelsalam A, Maestroni A, Seelam AJ, Ben Nasr M, Loretelli C, Mileto D, Rossi G, Pastore I, Montefusco L, Morpurgo PS, Plebani L, Rossi A, Chebat E, Bolla AM, Lunati ME, Mameli C, Macedoni M, Antinori S, Rusconi S, Gallieni M, Berra C, Folli F, Galli M, Gismondo MR, Zuccotti G, Fiorina P. Immunogenicity and Safety of SARS-CoV-2 mRNA Vaccines in a Cohort of Patients With Type 1 Diabetes. Diabetes. 2022 Aug 1;71(8):1800-1806. doi: 10.2337/db22-0053. PMID 35551366